CLINICAL TRIAL: NCT06735144
Title: A Multicenter, Open Label Phase I/II Clinical Study on the Safety, Tolerability, Pharmacokinetics, and Efficacy of FH-006 for Injection in Patients With Malignant Solid Tumors
Brief Title: Phase I/II Clinical Study of FH-006 for Injection in Patients With Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FH-006-101
Record Dates: First submitted 2024-12-06; First posted 2024-12-16 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2024-12

CONDITIONS: Malignant Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Queue A (Experimental)
  Interventions: Drug: FH-006
- Queue B (Experimental)
  Interventions: Drug: FH-006

INTERVENTIONS:
Drug: FH-006 — Intravenous injection once every two weeks (Q2W), with a treatment period of 28 days
  Arms: Queue A
Drug: FH-006 — administered once every 3 weeks (Q3W), with a treatment period of 21 days
  Arms: Queue B

SUMMARY:
Evaluate the safety, tolerability, pharmacokinetics, and immunogenicity of FH-006 in subjects with advanced malignant solid tumors, and determine the maximum tolerated dose (MTD) or maximum administered dose (MAD), recommended dose for phase II clinical trials (RP2D), and preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 to 75 (inclusive)
2. Subjects with histologically or cytologically confirmed recurrent or metastatic solid tumors who experience disease progression after standard treatment, or who do not have a standard treatment plan or are not suitable for standard treatment.
3. ECOG score is 0 or 1
4. An expected survival of ≥3 months
5. At least one target lesion according to RECIST v1.1 criteria
6. Has a good level of organ function
7. Patients voluntarily joined the study and signed informed consent

Exclusion Criteria:

1. Have other malignancies within the past 5 years
2. Active central nervous system metastasis without surgery or radiotherapy
3. Presence with uncontrollable third space effusion
4. Have undergone other anti-tumor treatment within 4 weeks before the first dose
5. Has severe infection within 4 weeks before the first medication
6. Any active autoimmune disease or a history of autoimmune disease
7. A history of immune deficiency
8. Has serious cardiovascular and cerebrovascular diseases
9. Clinically significant history of lung disease
10. The toxicity from previous anti-tumor treatment has not recovered to ≤ grade I
11. Having undergone surgery on important organs within 4 weeks prior to the first use of medication
12. Used attenuated live vaccine within 28 days prior to the first use of the investigational drug
13. Presence of other serious physical or mental diseases or laboratory abnormalities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
DLT: 21or28 days after the first administration of each subject | 21or28 days after the first administration of each subject
AE: from Day1 to 30 days after last dose | from Day1 to 30 days after last dose
Incidence and severity of serious adverse events (SAE): from Day1 to 30 days after last dose | from Day1 to 30 days after last dose
MTD or MAD： 21 or 28 days after the first dose of medication for each subject on dose escalation stage | 21 or 28 days after the first dose of medication for each subject on dose escalation stage
RP2D：Obtain two treatment evaluation data for the last subject during the dose expansion phase | Obtain two treatment evaluation data for the last subject during the dose expansion phase

SECONDARY OUTCOMES:
Immunogenic indicators: anti-FH-006 antibody (ADA) | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided